CLINICAL TRIAL: NCT05869851
Title: Comparison of Brace to Observation in Stable, Radiological Developmental Dysplasia of the Hip: A Multi-centre, International Randomized Controlled Non-inferiority Trial
Brief Title: Developmental Dysplasia of the Hip: Observation vs. Bracing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kishore Mulpuri, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H20-03750
Record Dates: First submitted 2023-05-10; First posted 2023-05-22 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Developmental Dysplasia of the Hip; Hip Dysplasia; Hip Dysplasia, Congenital; Hip Dysplasia, Developmental
MeSH Terms: conditions — Developmental Dysplasia of the Hip; Hip Dislocation; Hip Dislocation, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brace Treatment (Experimental): Patients randomized to the brace treatment group will be treated with a Pavlik harness for a minimum of six weeks.
  Interventions: Other: Pavlik Harness
- Active Monitoring (No Intervention): Patients randomized to the control group will undergo observation only.

INTERVENTIONS:
Other: Pavlik Harness — The Pavlik harness is an abduction brace used for treatment of hip dysplasia in infants. It keeps the hips in proper alignment to allow for appropriate growth and development of the joint.
  Arms: Brace Treatment

SUMMARY:
Developmental dysplasia of the hip (DDH) is the most common childhood hip condition. When caught early, bracing is the most frequently used treatment; however, the brace can disrupt important mother-baby bonding time in the newborn period and present challenges to daily living. In babies with mild DDH, some studies have suggested that their hips may improve naturally as they grow and develop. This study will look at whether careful monitoring can be just as good as bracing for babies diagnosed with mild DDH less than 3 months of age, potentially avoiding unnecessary treatment. This will be the first study to look at this question with babies being treated at different hospitals in seven different countries, so the results will make an impact on children and families worldwide.

DETAILED DESCRIPTION:
Early detection of developmental dysplasia of the hip (DDH) is critical to optimize outcomes and minimize long-term disability and impact on quality of life for the child and family. The burden of disease is significant, with a DDH diagnosis in 15-20/1000 live births. Even when treated, DDH is a leading cause of early hip replacement or development of osteoarthritis in young adults, with DDH reportedly accounting for 10-92% of all hip replacements. Consideration must also be given, however, to potential overtreatment of infants, particularly in more mild cases of hip instability or radiological dysplasia. The hip joint is immature during infancy, and many cases of mild-to-moderate DDH can spontaneously resolve as the hip joint matures through development. Brace treatment for approximately six weeks is common to address this radiological dysplasia; however, it is unclear whether this approach provides significant benefit above careful observation by ultrasound. While a conservative, less costly approach, brace treatment is not without potential complications and drawbacks. There are still substantial healthcare costs and resources associated with brace treatment, but there is potentially an under-recognized psychosocial cost in regard to preventing or disrupting mother-infant bonding in the newborn period. Coping with the difficulties of brace treatment can be stressful for families, particularly mothers of newborns, but the ultimate psychosocial impact has been under-researched to date. There is evidence to suggest that events occurring during establishment of breastfeeding may impact the mother's ability to breastfeed. The UK Hip Trial (2005) also found that maternal anxiety and worries about their infant's hip were increased with early brace treatment, but were not elevated by ultrasound monitoring in isolation. Further, bracing can present challenges to daily family life, including dressing, mobility, and the need for specialized furniture, car seats and other equipment. If observation alone is non-inferior to bracing for radiological dysplasia, unnecessary treatment may be avoided, potentially decreasing both the psychosocial impact of disrupted mother-infant bonding and needed healthcare resources and costs.

The investigators propose to utilize the existing collaborations and infrastructure of the Global Hip Dysplasia Registry (GHDR) and leverage their collaboration with a group in the Netherlands performing a similar Treatment with Active Monitoring (TRAM) trial to determine whether observation alone is sufficient for infants with clinically stable radiologically abnormal hips. Specifically, the investigators aim to:

1. Determine whether observation is non-inferior to bracing for infants with radiological dysplasia
2. Provide a strong recommendation for management of this subset of DDH patients
3. Compare findings to those of the Netherlands trial, which is being carried out in older patients (10-16 weeks at diagnosis)

This study will utilize the established infrastructure of the GHDR. GHDR was established in 2016, aimed at collecting longitudinal data on infants and children across the entire DDH spectrum. This specific trial will function as a targeted sub-study within the more extensive registry, and is a multi-centre, international prospective randomized non-inferiority trial designed to evaluate the necessity to treat infants with radiological hip dysplasia. In total, 14 of the centres currently contributing data to GHDR have agreed to participate and randomize eligible patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with radiological dysplasia of a clinically stable hip under three months (12 weeks) of age
* Radiological dysplasia will be defined as a centred hip with an alpha angle between 43 and 60 degrees and a percent coverage of the femoral head (FHC) greater than 35%, as measured on ultrasound exam

Exclusion Criteria:

* Patients presenting with radiological dysplasia older than three months (12 weeks) of age
* Patients presenting with clinical hip instability (Ortolani or Barlow positive)
* Patients with known or suspected neuromuscular, collagen, chromosomal or lower-extremity congenital abnormalities or syndromic-associated hip abnormalities
* Patients who received prior treatment (i.e. Pavlik harness) for DDH

Max Age: 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 514 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Acetabular Index | 2 years
  A measure of the steepness of the acetabular roof assessed on radiograph.

SECONDARY OUTCOMES:
Alpha Angle | 6 weeks
  This angle is measured via ultrasound and refers to the angle between the acetabular roof and vertical cortex of the ilium.
Beta Angle | 6 weeks
  This angle is measured via ultrasound and refers to the angle formed between the vertical cortex of the ilium and the triangular labral fibrocartilage (echogenic triangle).
Percent Femoral Head Coverage | 6 weeks
  Measured via ultrasound and assesses the percentage of the femoral epiphysis covered by the acetabular roof.
Number of Participants that Experienced Complications | 2 years
  Including development of femoral nerve palsy or avascular necrosis, progression of hip dysplasia, and need for further treatment.
Parent/Guardian Perception Questionnaire | 6 weeks
  A survey assessing parent/guardian perceptions of caring for and bonding with their child. Each question is scored on a 7-point likert scale from 3 (strongly agree) to -3 (strongly disagree) with total scores ranging from 33 to -33.
EuroQoL-5D | 6 weeks, 1 year, 2 years
  A survey assessing parent quality of life. Only the VAS portion of the questionnaire will be asked at each visit. The VAS is scored from 0 to 100 with higher scores indicating better health.
Parent/Guardian Satisfaction | 6 weeks, 1 year, 2 years
  Assessed using a VAS scored from 0 to 100 with higher scores indicating higher satisfaction.
Healthcare Resource Use Questionnaire | 6 weeks, 6 months, 1 year, 18 months, 2 years (Canadian centres only)
  Parent/guardian reported questionnaire to collect information about visits to health care professionals, imaging, medication use, additional treatments related to the diagnosis of DDH, and out of pocket costs.

OTHER OUTCOMES:
Centre Edge Angle | 5 years
  To be assessed for participants who elect to take part in the Global Hip Dysplasia Registry and have available data. Measured on x-ray, it is the angle formed between the vertical axis of the pelvis and a line from the centre of the femoral head to the lateral edge of the acetabulum.

CONTACTS AND LOCATIONS:
Overall Officials: Kishore Mulpuri, FRCSC, Principal Investigator — University of British Columbia; Emily Schaeffer, PhD, Study Director — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
While we will not make individual participant data available for this study, we do intend to disseminate study results to participants, researchers and the broader public.
  Our team works closely with patient partners, healthcare personnel, our collaborators and the broader medical/scientific community to determine appropriate ways to disseminate study results. We intend to prepare plain language summaries and visual/video abstracts of study results, which will be emailed to participants (those whom provided consent for email contact). These visual abstracts will also be posted to our lab's social media accounts, as well as that of our supporter, the I'm a HIPpy Foundation, who works closely with our patient and family community.

REFERENCES:
- [Derived] Zomar BO, Bone JN, Nguyen V, Mulpuri K, Kelley S; GHD Study Group; Schaeffer EK. Comparison of brace to observation in stable, radiological developmental dysplasia of the hip: a protocol for a global multicentre non-inferiority randomised trial. BMJ Open. 2024 Jul 8;14(7):e084738. doi: 10.1136/bmjopen-2024-084738. PMID 38977361